CLINICAL TRIAL: NCT02367469
Title: Tryptophan Metabolism in Human Brain Tumors
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Csaba Juhasz, Principal Investigator, Wayne State University
Other Study IDs: NCI Tryptophan; CA123451 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2015-02-12; First posted 2015-02-20 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Brain Tumors
Keywords: recurrent brain tumors; brain tumors; Newly diagnosed brain tumors
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will collect and analyze tumor specimens obtained after AMT-PET during tumor resection (if not used for routine histopathology). Various histopathologic features will be studied, e.g., tumor proliferative activity, expression of amino acid transporter as well as enzymes and metabolites of the kynurenine pathway, and these will also be correlated with neuroimaging findings.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brain Tumors: Patients with newly diagnosed or recurrent brain tumors will be studied.

SUMMARY:
The main purpose of this study is to determine the potential clinical utility of PET imaging using the radiotracer [C-11]alpha-methyl-L-tryptophan in the diagnosis, differentiation and monitoring of various brain tumors, both before and after initial treatment. We will also study mechanisms and clinical significance of abnormal brain tumor tryptophan metabolism using resected tumor tissues.

DETAILED DESCRIPTION:
If you agree to take part in this research study, you will be asked to have:

1. a PET scan, 2. brief clinical questionnaires, and 3. biochemical studies of blood and tumor tissue. You may also have a second PET scan later, if you undergo therapy (such as surgery and/or brain radiation), to determine if there are PET signs of tumor. Your ability to participate in the study will be based, in part, on the results of the magnetic resonance images (MRI) in your medical chart from earlier clinical procedures. Once we receive the results of the PET scan, these will be compared to the MRI in order to help us analyze whether the tryptophan uptake tells us anything about the type of tumor in your brain. It will take about 3 hours to complete the PET scan; this includes the completion of the questionnaires, preparation and scanning. The actual scanning time will be 70 minutes. If you are a female of child-bearing age, we will need a small urine sample from you before starting the PET scanning procedure to make absolutely sure that you do not have unknown pregnancy for which radiation exposure might be harmful.

1. The PET scan will be used to measure the accumulation of the injected radioactive tracer AMT in your brain. To make this measurement more accurate, we will use your clinically obtained MRI scan(s), which was used to diagnose the tumor, to identify the exact location and extent of the tumor. For the PET scan, an intravenous catheter (a small tube placed in your vein) will be inserted for the injection of the AMT for this PET scan. It is the tracer that the PET scanner "sees" when performing the scan. The amount of the tracer, which will be given is very small (5 ml, the volume of a teaspoon), and therefore no side effects are expected from the tracer itself. A second intravenous catheter will be inserted to collect blood samples during the scan; a total of less than 2 teaspoons of blood will be collected. Participants may be sedated (put into sleep with some medicine) if they are unable to remain still for the scanning period.
2. On the day of the PET scan, we will ask you to fill out a brief clinical questionnaire, and also an additional multiple-choice questionnaire to screen for potential mood problems (which often coincide with brain tumors). Participants with a potential speech (comprehension) problem will also be administered a brief speech test. The goal of these tests is to identify various clinical problems that can be associated with brain tumors and affected by abnormal tryptophan metabolism that we measure with the PET scan.
3. If you have surgery to remove the tumor, a portion of the removed tissue will be used for biochemical studies. The doctor will not remove more tissue than needed for your care. The blood (obtained during the PET scanning) and tumor tissue (obtained during surgery) will be processed for analysis and stored in a locked container or freezer in a laboratory. In addition, we will review the clinical pathology report, so that we can correlate your PET results to type and grade of the tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical and MRI diagnosis of an intracranial lesion suspicious for a brain tumor, including primary and metastatic tumors, or a possible residual or recurrent brain tumor (based on clinical imaging); or history of glioma treatment with chemoradiation, even if no definite progression is found on clinical MRI.
2. Age ≥13 years.

Exclusion Criteria:

1. Severe increased intracranial pressure, status epilepticus, or other symptoms requiring emergency or urgent intervention.
2. Resective surgery within 2 months prior to the PET scan (acute/subacute post-surgical inflammatory changes may cause false positive increases on AMT PET).
3. Positive pregnancy test (because of radiation involved in PET scanning).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed or recurrent brain tumors will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
In newly diagnosed tumors | single time-point
  Diagnostic accuracy of AMT-PET to differentiate brain tumor types and detect tumor infiltration of the brain.
In previously treated tumors | single time-point
  Accuracy of AMT-PET to predict post-treatment progression and differentiate recurrent tumors from radiation-induced changes, as compared to clinical MRI.

SECONDARY OUTCOMES:
Tryptophan metabolism | single time-point
  To evaluate activity of the kynurenine pathway of tryptophan metabolism in resected tumor tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Csaba Juhasz, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jeong JW, Lee MH, John F, Robinette NL, Amit-Yousif AJ, Barger GR, Mittal S, Juhasz C. Feasibility of Multimodal MRI-Based Deep Learning Prediction of High Amino Acid Uptake Regions and Survival in Patients With Glioblastoma. Front Neurol. 2019 Dec 17;10:1305. doi: 10.3389/fneur.2019.01305. eCollection 2019. PMID 31920928
- [Result] John F, Robinette NL, Amit-Yousif AJ, Bosnyak E, Barger GR, Shah KD, Mittal S, Juhasz C. Multimodal Imaging of Nonenhancing Glioblastoma Regions. Mol Imaging. 2019 Jan-Dec;18:1536012119885222. doi: 10.1177/1536012119885222. PMID 31736437
- [Result] John F, Bosnyak E, Robinette NL, Amit-Yousif AJ, Barger GR, Shah KD, Michelhaugh SK, Klinger NV, Mittal S, Juhasz C. Multimodal imaging-defined subregions in newly diagnosed glioblastoma: impact on overall survival. Neuro Oncol. 2019 Feb 14;21(2):264-273. doi: 10.1093/neuonc/noy169. PMID 30346623
- [Result] Guastella AR, Michelhaugh SK, Klinger NV, Fadel HA, Kiousis S, Ali-Fehmi R, Kupsky WJ, Juhasz C, Mittal S. Investigation of the aryl hydrocarbon receptor and the intrinsic tumoral component of the kynurenine pathway of tryptophan metabolism in primary brain tumors. J Neurooncol. 2018 Sep;139(2):239-249. doi: 10.1007/s11060-018-2869-6. Epub 2018 Apr 17. PMID 29667084
- [Result] Bosnyak E, Michelhaugh SK, Klinger NV, Kamson DO, Barger GR, Mittal S, Juhasz C. Prognostic Molecular and Imaging Biomarkers in Primary Glioblastoma. Clin Nucl Med. 2017 May;42(5):341-347. doi: 10.1097/RLU.0000000000001577. PMID 28195901
- [Result] Bosnyak E, Kamson DO, Robinette NL, Barger GR, Mittal S, Juhasz C. Tryptophan PET predicts spatial and temporal patterns of post-treatment glioblastoma progression detected by contrast-enhanced MRI. J Neurooncol. 2016 Jan;126(2):317-25. doi: 10.1007/s11060-015-1970-3. Epub 2015 Oct 29. PMID 26514361
- [Result] Bosnyak E, Kamson DO, Behen ME, Barger GR, Mittal S, Juhasz C. Imaging cerebral tryptophan metabolism in brain tumor-associated depression. EJNMMI Res. 2015 Dec;5(1):56. doi: 10.1186/s13550-015-0136-9. Epub 2015 Oct 17. PMID 26475140
- [Result] Jeong JW, Juhasz C, Mittal S, Bosnyak E, Kamson DO, Barger GR, Robinette NL, Kupsky WJ, Chugani DC. Multi-modal imaging of tumor cellularity and Tryptophan metabolism in human Gliomas. Cancer Imaging. 2015 Aug 6;15(1):10. doi: 10.1186/s40644-015-0045-1. PMID 26245742
- [Result] John F, Michelhaugh SK, Barger GR, Mittal S, Juhasz C. Depression and tryptophan metabolism in patients with primary brain tumors: Clinical and molecular imaging correlates. Brain Imaging Behav. 2021 Apr;15(2):974-985. doi: 10.1007/s11682-020-00305-7. PMID 32767048